CLINICAL TRIAL: NCT05670418
Title: Cognitive Function Analysis and qEEG Study in Long COVID-19 Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr Yetty Ramli SpS, Medical Staff & Lecturer, Indonesia University
Other Study IDs: 22-05-0578
Record Dates: First submitted 2022-11-22; First posted 2023-01-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Long COVID-19 Syndrome
Keywords: Long COVID-19 Syndrome; COVID-19; Quantitative electroencephalography; Case-control study
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long COVID-19: Patients post-COVID-19 with Long COVID-19 Syndrome
  Interventions: Device: Quantitative Electroencephalography
- COVID-19: Patients post-COVID-19 without Long COVID-19 Syndrome
  Interventions: Device: Quantitative Electroencephalography

INTERVENTIONS:
Device: Quantitative Electroencephalography — Each qEEG examination of one person lasted about 20 minutes and included two stages: the first-recording of brain waves with eyes closed (5 min), the other with eyes open (5 min)

SUMMARY:
Over than 30% individuals with COVID-19, including the asymptomatic ones, and around 80% of patients hospitalized with COVID-19 may experience post-COVID sequelae, which is commonly referred to as Long COVID Syndrome. This condition has ties to decreased cognitive function and may lead to neuropsychiatric disorders but still need to be studied further. Using a cross-sectional design, this study will analyze the relationship between cognitive function and neuropsychiatric disorders with brain wave activity in Long COVID patients.

The investigators conducted assessments utilizing the quantitative electroencephalogram (qEEG) measurement method and interviews using instruments such as the MOCA questionnaire and Self Rating Questionnaire (SRQ). With this qEEG examination, the investigators hoped that there will be an imbalance/abnormality of brain wave activity that arises related to impaired cognitive function.

DETAILED DESCRIPTION:
This study is aimed to analyze the cognitive function and neuropsychiatry disorders with brain wave activity using qEEG that occurs after COVID/Long Covid Syndrome.

The whole procedure will run for approximately 12 weeks based on the long COVID range.

The determinants of long COVID patients include: never been vaccinated, old age, comorbid, female population, and hospitalized patients.

The total number of subjects with the post-COVID syndrome in the proportion test is 30 subjects.

The measuring instruments used to measure the decline in cognitive function are the MOCA questionnaire and Self Rating Questionnaire (SRQ).

The target population is post-COVID-19 patients with Long COVID Syndrome.

The accessible population is post-COVID-19 patients who have been treated at RSCM Kiara and have regular checkups at the RSCM polyclinic with Long COVID Syndrome for 12 weeks or more.

The control population is post-COVID-19 patients who managed to recover without symptoms.

The Long COVID Syndrome patients who meet the inclusion criteria and have signed the consent.

ELIGIBILITY:
Inclusion Criteria:

1. Post-COVID-19 patients with Long COVID-19 Syndrome
2. Over 18 years old
3. Willing to participate in the research
4. Completed the Montreal Cognitive Assessment (MoCA) and Self Rating Questionnaire (SRQ)

Exclusion Criteria:

1. Patients with neuropsychiatric disorders before being infected with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 Patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Through study completion, an average of 1 year
  Cognitive Function will be assessed using the qEEG, with an abnormality of brain wave activity, it indicates impairment of cognitive function

SECONDARY OUTCOMES:
Cognitive quality Assessed by MOCA | Through study completion, an average of 1 year
  Severe score: ≤10 Moderate score: 10-17 Mild score: 18-25 Normal score: 26-30
Self Rating Questionnaire (SRQ) | Through study completion, an average of 1 year
  Lowest score: 0 Highest score: 20. Higher score indicates better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Manunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia